CLINICAL TRIAL: NCT03017456
Title: Prostate Cancer Survivorship 360°
Brief Title: PC 360 Survivorship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Vancouver Prostate Centre (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15-5045-CE
Record Dates: First submitted 2017-01-04; First posted 2017-01-11 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
Keywords: Survivorship; Prostate Cancer; Survivorship Care Plan
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (UC) (No Intervention): Patients in the UC arm will not receive the study intervention (behavioral) and instead will receive care according to usual practice. This usually involves a brief office visit (approximately 5-10 minutes) with pertinent history and physical examination related to surgical/radiation recovery, review of the pathology and general instructions regarding the next step in follow-up.
- SCP-Intervention vs usual care (Active Comparator): behavioral intervention vs control Patients in the SCP-Int arm will be asked to attend a one-time appointment with a trained oncology nurse. The SCP-Int is comprised of a 30-minute nurse-led face-to-face intervention and the provision of a tailored PC-specific SCP (PC-SCP). Persistent effects and concerns that are identified will prompt the development of a tailored management plan captured within the PC-SCP. Relevant patient education materials will be linked electronically. Nurses will use motivational interviewing techniques to effective in increase healthy behaviors and empower the PC survivor to actively self-manage persistent treatment effects and to decrease their risk of late effects by providing effective health information, support, and self-management support.
  Interventions: Behavioral: Survivorship Care Plan

INTERVENTIONS:
Behavioral: Survivorship Care Plan — SCP-Intervention: Patients in the SCP-Int arm will attend a one-time appointment with a trained oncology nurse while the patients in the UC arm will receive care according to the hospital standards for follow-up care. The intervention will be delivered during a regular follow-up appointment, face-to-face and will inform and educate patients on self-management and support as well as promote access to and coordination of post-treatment care. The appointment will focus on empowering the PC survivor to actively self-manage persistent treatment effects and to decrease their risk of late effects by providing effective health information, support, and self-management support. Nurses will integrate a number of "active behavior change ingredients" including the integration of motivational interviewing techniques which are effective in increasing healthy behaviors.
  Other Names: PC 360-SCP
  Arms: SCP-Intervention vs usual care

SUMMARY:
Prostate Cancer Survivorship 360º is a collaboration-based initiative involving prostate cancer (PC) and survivorship researchers/clinicians from three Canadian prostate centers with the goal of identifying and tracking unmet supportive care needs of patients with localized PC and responding to these needs through survivorship care. The current randomized control trail (RCT) will focus on the development and evaluation of a facilitated electronic Prostate Cancer Survivorship Care Plan (PC-SCP). The aims of this project are: 1) to develop an appropriate and tailored SCP and transition care delivery process; and 2) to conduct an RCT to evaluate whether a personalized PC SCP intervention is more effective than usual care (UC) on patient activation (primary outcome) and access to services, self-Management support, satisfaction with information, HRQoL and cancer worry (secondary outcomes). Data from a multi-site prospective database- Prostate Cancer Survivorship Information System (PC360-IS) will be used to electronically populate the survivorship care plans. Overall, this proposal represents initial steps in uniting the country in sharing programmatic resources, data, expertise, and enthusiasm to transform survivorship care for men with PC and their families.

DETAILED DESCRIPTION:
A Phase III RCT will evaluate the superiority of a Survivorship Care Plan (SCP) intervention (SCP-Int) compared with usual care (UC) after primary curative prostate cancer (PC) treatment. Each of the three sites has designated clinical study leads (AM, LG, and ST), high referral volumes and study leads' patients will be entered into the PC360-IS database which will be interfaced to the PC-SCP system to consolidate patient details and generate personalized SCPs. Research ethics approval will be obtained at each site. The trial will be registered with clinicaltrials.gov and reported using the CONSORT recommendations for trials.

The study population inclusion criteria are as follows: Histologically confirmed localized (T1-T3N0M0) PC; age at diagnosis >18 years; treated with curative intent; treatment received >1 month and <6 months; disease-free as defined by absence of somatic disease activity parameters as per oncologist/urologist; consented to participate in the PC360-IS database. Exclusion Criteria: Patients who do not receive treatment and are followed by active surveillance; inability to complete study questionnaires.

Eligible patients will be randomly assigned to either the intervention arm or the control arm. A biostatistician will randomly assign participants to ensure that both the study RA and the participants are unaware of the treatment (SCP-int)/control groups (UC). Consenting patients will be registered into the study and randomized to receive either the SCP-Int or UC. Patients in the SCP-Int arm will be scheduled for the SCP-Int appointment on the same day as the patient's first (or second) follow-up appointment.

Eligible patients will be sent a study information letter which will be signed by the patient's urologist/ oncologist one month after the end of primary treatment. The RA will then contact patients to further explain the study. If agreeable, the patients will be sent consent forms, two stamped envelopes, and a baseline questionnaire to complete prior to the scheduled follow-up appointment. The patients will be asked to mail back the signed consent form and the completed questionnaire in each the envelopes provided.

Participants will have as much time as needed to decide if the participants would like to participate in the study prior to signing the consent form. The Research Analyst will obtain consent.

Planned trial interventions: SCP-Int: Patients in the SCP-Int arm will be asked to attend a one-time appointment with a trained oncology nurse (study nurse). To avoid additional travel and related costs to the patient, this appointment will be scheduled on the same day as the patient's follow-up appointment. The SCP-Int is comprised of two components: a 30-minute nurse-led face-to-face intervention and the provision of a tailored PC-specific SCP (PC-SCP). The intervention will be developed based on an established person-centred nursing framework with a tailored approach to customizing the intervention to the individual and will focus on the provision of self-management education and support and promote access to and coordination of post-treatment care including appropriate referrals to relevant programs and services (including TrueNTH solutions). The content of the PC-SCP will provide structure to the appointment. Persistent effects and concerns that are identified will prompt the development of a tailored management plan (i.e. patient education, referral to programs and services) captured within the PC-SCP. Relevant patient education and TrueNTH materials will be linked electronically. The appointment will focus on empowering the PC survivor to actively self-manage persistent treatment effects and to decrease the patients' risk of late effects by providing effective health information, support, and self-management support. Nurses will integrate a number of "active behaviour change ingredients" including the integration of motivational interviewing techniques which are effective in increasing healthy behaviours. Usual Care (UC): Patients in the UC arm will receive care according to usual practice. This usually involves a brief office visit (approximately 5-10 minutes) with pertinent history and physical examination related to surgical/radiation recovery, review of the pathology and general instructions regarding the next step in follow-up. In addition, patients in the UC arm will be able to access any supportive care programs or service available at the hospital according to usual practice. Currently, SCPs and dedicated transition appointments are not provided as part of a standard of care.

Allocation to trial groups: Patients will be allocated to either SCP-Int or UC by the Department of Biostatistics at Princess Margaret using a computer-generated randomization process (random blocks known only to statisticians). The research coordinator will telephone Biostatistics staff, who will not be involved in recruitment, to obtain the subject's assignment. Eligible patients from each site will be approached until the target number of participants is reached (or until a decision is made to stop recruitment).

Data collection: Data will be collected and analyzed according to the outlined project aims. Based on CONSORT criteria, a screening log will enable data collection on eligible and non-recruited patients with reasons for non-recruitment recorded when known. All data will be entered into a secured, password protected database within the UHN server. A separate database will be used for participant tracking to prevent re-approaching patients unnecessarily, and to ensure patients are receiving the questionnaire packages according to the study timeline.

Proposed primary and secondary outcome measures:

The outcome measures were chosen based on recent consensus and recommendations on the evaluation of SCPs. Patients will be assessed at baseline (T0), 6 (T1), and 12 (T2) months post-treatment. This questionnaire package is estimated to take 45 minutes to complete.

Primary Outcome: Patient activation will be measured using the Patient Activation Measure (PAM-13), a 13-items measure assessing knowledge, skills, beliefs, and confidence in managing health and health care. Patient activation is strongly related to a broad range of health-related outcomes. The primary outcome will be the overall score of the 13 items collected at T2.

Secondary Outcomes: a) Supportive care services utilization: using the Health and Social Services Utilization Inventory (HSSUI) modified for use in cancer populations. Service types are grouped into five categories: Health Professionals, Institutional/Hospital Programs; Nursing and Homemaker Support Programs; Other Community and Social Support Program/Resources (will include True NTH solutions); Programs/Resources.; b) Self-Management Support will be assessed using the Health Education Impact Questionnaire (heiQ), designed to evaluate outcomes from patient education and self-management interventions for people with chronic conditions; c) Satisfaction with Information will be measured with the 25-item European Organisation for Research and Treatment of Cancer Quality of Life INFO25 module which evaluates satisfaction with information received by cancer patients; d) Quality of Life will be measured using the Expanded Prostate Cancer Index Composite (EPIC) which assesses PC-specific quality of life, and e) Cancer Worry will be measured using the Assessment of Survivors Concerns (ASC) measure which assesses fear of recurrence and health in cancer survivors.

Proposed sample size and justification: Our sample size calculations are based on 85% power with an alpha-level of 0.05, a standard deviation of 16 and a difference between groups of 8 points on the primary outcome (or half a standard deviation difference). Given these specifications, the required sample size is 146 patients (or 73 patients per arm). Assuming attrition of up to 20%, 180 patients will be recruited (or 90 patients per arm). Based on previous studies, we expect to enroll about 70% of eligible patients. The number of potentially eligible patients from participating sites is estimated to vary between 15-30 patients per month. Based on these estimates and our anticipated participation rates, we anticipate recruiting 20 patients per month with total recruitment completed within 9 months. We anticipate at least 80% will complete the 12-month post-treatment follow-up. We will use multiple strategies to promote retention and prevent attrition. Reasons for participant attrition will be documented.

Proposed analyses: Analyses will be performed adhering to the intention to treat principle. Descriptive statistics will be used to summarize baseline demographic and clinical characteristics of participants in both groups. Recruitment bias and possible differential attrition will be assessed by calculating the standardized differences between the two arms. The overall PAM-13 score at 12 months adjusted for the baseline score will be compared between the two arms using the t-test if the data appears normal or the Mann-Whitney test otherwise. A p-value<=0.05 will be deemed significant. Secondary analyses of all scores at each time point will be conducted utilizing the mixed effect modeling to account for the intra-patient and intra-centre dependency due to the repeated measures within a patient and the multi-centre design. The residuals will be inspected and data will be transformed when necessary. Due to multiple testing for the secondary analyses a Hochberg-Benjamini approach will be used to ensure that the type I error rate does not exceed 0.05.

Cost-utility analyses: The analysis will also include a trial-based cost utility analysis. The health utility measured using the PORPUS-U and EQ-5D instruments will be used to provide patient-specific and group-mean estimates of quality-adjusted survival (Quality Adjusted Life Years). Costs from the payer perspective and from the societal perspective will be gathered using the HSSUI and an estimate of intervention costs. Inverse probability weighting will be used to adjust for induced dependent censoring. A net benefit regression approach will be employed to explore predictors of cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed localized (T1-T3N0M0) PC
* age at diagnosis >18 years
* treated with curative intent
* treatment received >1 month and <6 months
* disease-free as defined by absence of somatic disease activity parameters as per oncologist/urologist
* consented to participate in the PC360-IS database.

Exclusion Criteria:

* Patients who do not receive treatment and are followed by active surveillance
* inability to complete study questionnaires.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in the Patient Activation measure questionnaire | Change from baseline (prior to intervention), 6 months post intervention, 12 months post intervention.

SECONDARY OUTCOMES:
Changes in the Health and Social Services Utilization Inventory | change from baseline (prior to intervention), 6 months post intervention, 12 months post intervention.
Changes in the Health Education Impact Questionnaire | Change from baseline (prior to intervention), 6 months post intervention, 12 months post intervention.
Changes in the Quality of Life INFO25 module | Change from baseline (prior to intervention), 6 months post intervention, 12 months post intervention.
Changes in the Expanded Prostate Cancer Index Composite | Change from baseline (prior to intervention), 6 months post intervention, 12 months post intervention.
Changes in the Assessment of Survivors Concerns measure | baseline (prior to intervention), 6 months post intervention, 12 months post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Jones, PhD, Principal Investigator — Princess Margaret Cancer Centre, University Health Network
Locations (3):
- Canada (3):
  - Vancouver Prostate Centre, Vancouver, British Columbia
  - University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones JM, Matthew A, Tanguay S, Higano CS, Goldenberg L, Howell D, Maganti M. A Tailored Electronic Survivorship Care Plan for Prostate Cancer Survivors: A Multicenter Randomized Controlled Trial. J Urol. 2025 Apr;213(4):407-416. doi: 10.1097/JU.0000000000004359. Epub 2024 Dec 20. PMID 39705576